CLINICAL TRIAL: NCT02057419
Title: K24: Advancing Reproductive Health: Women's Input on Sexual Health (Project WISH)
Brief Title: Women's Input on Sexual Health
Acronym: WISH
Status: Completed | Type: Observational
Sponsor: The Miriam Hospital (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: TMH-506070; K24HD062645 (NIH)
Record Dates: First submitted 2014-01-31; First posted 2014-02-07 (Estimated); Results first posted 2025-10-24 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Intravaginal Ring Use
Keywords: contraception; contraceptive methods; user experience

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Intravaginal Ring Users: Use IVR for 3-month period and report user sensory perceptions and experiences.

SUMMARY:
The purpose of this study is to answer the following question: How do user sensory perceptions and experiences (USPEs) for IVRS differ between initial and continued use and how can this knowledge help product developers better understand how to design new IVR products and develop behavioral (or point-of-care) interventions to optimize use?

DETAILED DESCRIPTION:
Background: Sexual and reproductive health (SRH) is a global public health priority. Providing efficacious SRH technologies that have the greatest likelihood of use will have the greatest impact on women's health. Critical to use is "acceptability." However, current conceptualizations of adherence and acceptability fail to fully articulate and account for the user experience. Given the recent development of various IVR technologies and the potential for multipurpose technologies, the impact on global public health would be far-reaching, affecting reproductive health in women and men: decreasing STI incidence, minimizing unplanned pregnancies, and decreasing morbidity and mortality due to a range of other reproductive health conditions.

Condition: Participants will use an IVR for a period of three months and report sensory perceptions and use experiences.

Methodology and Data Collection: Volunteers (N~6-10) will first be screened for the study using a brief questionnaire. Those who are interested in contraception and are eligible based on their responses to the prescreen will then complete a clinical screening visit and pregnancy test. Once enrolled participants will complete a survey that asks questions about demographics and sexual and reproductive history.

During the course of the study, participants will evaluate their use of an IVR. IVRs will be used for three consecutive months. They will be given a three-month supply of the product at the beginning of the use period. About once a month, each participant will be required to complete a web survey about their experience with the study product.

All participants complete a final survey that will ask about their experiences with the study product.

ELIGIBILITY:
Inclusion Criteria:

* are between the ages of 18 and 45 at prescreening,
* report vaginal sex with a man in the past month at prescreening,
* are not pregnant (self-report, confirmed at V1, V2, and V3 by urine HcG test) and report no intention to become pregnant during the course of the study,
* report negative or unknown HIV status,
* report a need for contraceptive products and
* are willing and able to provide informed consent.

Exclusion Criteria:

* self-report pregnancy, have a positive urine pregnancy test at Visits 1, 2, or 3, or intend to become pregnant during the course of the study,
* self-report breast feeding,
* self-report a vaginal delivery or other reproductive surgical procedure in the past 30 days,
* self-report being HIV-positive,
* self-report being diagnosed with or having an active sexually transmitted infection (STI) in the past 12 months,
* self-report an allergy or sensitivity to any of the study products,
* do not have a cell phone or internet access,
* are unable or unwilling to give informed consent, or
* have any condition that, in the opinion of the study clinician(s) or principle investigator, would compromise the participant's ability to participate in the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Females who are 18-45 years old, HIV negative or unknown (self report), non-pregnant (urine test) and not intending to get pregnant (self-report), report vaginal sex with a man in the past month, and present with a need/desire for contraception.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2014-04-14 (Actual); Primary Completion 2016-06-24 (Actual); Study Completion 2018-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kate Guthrie, PhD, Principal Investigator — The Miriam Hospital: Centers for Behavioral & Preventive Medicine
Locations (1):
- The Miriam Hospital: Centers for Behavioral & Preventive Medicine, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited (RI, MA USA) via call-lists, flyers, ads, internet/social media, clinics, CBOs, word-of-mouth.
Period: Overall Study
Arm/Group | Intravaginal Ring Users
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Female participants using IVR for a period of 3 months
Arm/Group | Intravaginal Ring Users
Number analyzed (Participants) | 8
Age, Customized [Count of Participants; unit: Participants]
  18-29 | 6
  30-45 | 2
Sex/Gender, Customized [Number; unit: participants]
  Female | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Latina or Hispanic | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8
Marital Status [Count of Participants; unit: Participants]
  Never Married | 7
  Married | 0
  Separated | 0
  Divorced | 1
  Widowed | 0
Yearly Income [Count of Participants; unit: Participants]
  Less than $15,000 a year | 0
  $15,000 to $36,000 a year | 6
  $36,000 or more a year | 2
Health Insurance Coverage [Count of Participants; unit: Participants]
  Through a current or former employer or union | 4
  Purchased directly from an insurance company | 1
  Medicare due to a disability | 0
  Medicaid, medical assistance, or other kind of government assistance plan | 0
  TRICARE or other military health care | 0
  Covered by VA healthcare | 0
  Covered by the Indian Health Service | 0
  Another kind of health care insurance or health coverage plan_Parents' Insurance | 1
  Currently do not have health insurance | 2
Typical Tampon Use [Count of Participants; unit: Participants]
  Yes | 5
  No | 3

OUTCOME MEASURES:

1. Primary Outcome: USPE Scale Scores
Description: User sensory perceptions and experiences (USPEs) with the IVR will be captured approximately monthly over a 90 day use period. USPE Sum of averaged item means/# items (min:max 1:5); 1=Do not agree at all;2=Agree a little;3=Agree somewhat;4=Agree a lot;5=Agree completely.
  Product: IVR
  USPE Scales: Initial Penetration and First Strokes: Smoothness/lubricity; Awareness: Feel (not) intravaginally during sex; Discharge Look: Appearance of discharge; Discharge: Sensations of discharge during and after sex inside and outside body; Pleasure: Participant and partner's stimulation
  A higher score indicates greater agreement with subscale characteristics being reported on.
Time Frame: Up to 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intravaginal Ring Users
Number analyzed (Participants) | 8
score on a scale
  Initial Penetration & First Strokes (Month 1 IVR) | 3.73 (1.55)
  Initial Penetration & First Strokes (Month 3 IVR) | 3.63 (1.21)
  Discharge (Month 1 IVR) | 1.85 (1.41)
  Discharge (Month 3 IVR) | 2.02 (1.49)
  Discharge Look (Month 1 IVR) | 3.13 (1.58)
  Discharge Look (Month 3 IVR) | 3.07 (1.59)
  Awareness (Month 1 IVR) | 1.84 (0.86)
  Awareness (Month 3 IVR) | 1.82 (1.02)
  Pleasure (Month 1 IVR) | 1.63 (0.63)
  Pleasure (Month 3 IVR) | 2.81 (1.12)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Intravaginal Ring Users
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 2/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravaginal Ring Users (N=8)
Increased Vaginal Discharge (Reproductive system and breast disorders) | 1 (1) — Ppt noticed thick white chunks in her vagina when she went to feel for the ring. There was no odor and no other symptoms. Pt saw her PCP about a week and a half after the onset of symptoms. PCP believes chunks were not related to IVR use.
Tooth Infection (Infections and infestations) | 1 (1) — Pt noted during final visit after completion of 3-month use of IVR that she saw her PCP regarding a tooth infection. Pt was prescribed antibiotics and made plan for tooth extraction. Pt's symptoms did not affect her participation in the study.

LIMITATIONS AND CAVEATS:
User Sensory Perceptions & Experience (USPE) scales adapted and were used for the first time to evaluate IVR use in Project WISH.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No